CLINICAL TRIAL: NCT03111017
Title: Mechanisms and Management of Exercise Intolerance in Older Heart Failure Patients With Preserved Ejection Fraction
Brief Title: Mechanisms and Management of Exercise Intolerance in Older Heart Failure Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas at Arlington (Other)
Responsible Party: Principal Investigator, Mark Haykowsky, Professor & Moritz Chair in Geriatrics, College of Nursing and Health Innovation, The University of Texas at Arlington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 1R15NR016826-01 (NIH)
Record Dates: First submitted 2017-03-25; First posted 2017-04-12 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure, Diastolic
Keywords: muscle sympathetic nerve activity; exercise tolerance; exercise training; peak oxygen uptake
MeSH Terms: conditions — Heart Failure, Diastolic | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Training (Experimental): Subjects will perform continuous endurance exercise (arm and leg cycle on Schwinn AD6 Airdyne ergometer, treadmill walking) 3 days per week. During the first 4-weeks, the exercise intensity will be set at 60%-70% of heart rate reserve and will increase by 5% per month. The initial exercise duration be 30 minutes and will gradually increase by 10 minutes every month. A 5-minute warm up and cool-down will precede and follow the aerobic conditioning phase. After the aerobic training phase is completed, patients will also perform unilateral handgrip exercise at an initial intensity of 50% maximal voluntary contraction for 1 set of 10 repetitions, and the intensity and sets will increase by 5% and 1 set, respectively each month.
  Interventions: Other: Exercise Training
- Attention Control (No Intervention): These subjects will be asked to continue with normal activity and will not be given any exercise training. The subjects will be contacted by the study coordinator at pre-arranged times and dates once a month and involve inquiry regarding overall well-being of the subject.

INTERVENTIONS:
Other: Exercise Training — HFpEF patients randomized to either 16 weeks of exercise training or attention control group.
  Arms: Exercise Training

SUMMARY:
Heart failure with preserved ejection fraction (HFpEF) is the fastest growing form of heart failure with a high morbidity and mortality rate, and is associated with severe exercise intolerance. The mechanisms responsible for the reduced exercise tolerance remain poorly understood. The investigators propose a novel paradigm shift, focusing on peripheral limitations to exercise. In particular, the investigators will test the hypothesis that muscle sympathetic nerve activity (MSNA) is elevated in older HFpEF patients compared to healthy controls, and is associated with reduced exercise tolerance. The investigators will also test whether 16-weeks of exercise training will lower MSNA compared to attention control, and correlate with improved exercise tolerance in older HFpEF patients.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction is the fastest growing form of heart failure, is almost exclusively found in older persons, particularly older women, and is associated with a high morbidity and mortality rate. The primary chronic symptom in HFpEF patients is severe exercise intolerance measured objectively as decreased peak exercise oxygen uptake (peak VO2). A consequence of the reduced exercise tolerance is that activities of daily living require near maximal effort, resulting in further deconditioning and reduced quality of life. The majority of work to date has focused on cardiac limitations, showing impaired cardiac output and marked diastolic dysfunction. Although these findings have provided important insight into the pathophysiology of HFpEF, drug therapies targeting cardiac function do not improve peak VO2, quality of life, or survival in HFpEF patients.

Older HFpEF patients have multiple skeletal muscle abnormalities including reduced skeletal muscle oxidative capacity and capillary-to-fiber ratio resulting in increased anaerobic metabolism during low-level exercise. Importantly, accumulation of anaerobic metabolites within the exercising muscles are known to activate skeletal muscle afferent fibers (called metaboreceptors), that elicit a reflex-mediated increase in efferent muscle sympathetic (vasoconstrictor) nerve activity (MSNA). The investigators here propose a novel paradigm of exercise intolerance in older HFpEF patients whereby skeletal muscle abnormalities lead to overactivation of the muscle metaboreflex and MSNA mediated vasoconstriction that limits delivery of oxygenated blood to the active muscles. Further, exercise training mediated improvements in skeletal muscle function will alleviate the metaboreflex, thereby reducing MSNA and improve oxygen delivery to the contracting muscles.

To test this novel paradigm, the investigators will first perform an initial cross-sectional comparison of older (≥60 years) HFpEF patients (N=24) with age and sex-matched healthy controls (N=24), and then enter the HFpEF patients into a randomized, controlled, single blind, trial of exercise training to test the following hypothesis: (i) that MSNA is elevated in older HFpEF patients compared to healthy controls, and is associated with reduced peak VO2, physical functional performance, aerobic endurance, muscle blood flow, and quality of life; and (ii) Exercise training will attenuate MSNA compared to attention control, and will correlate with improved peak VO2, physical functional performance, aerobic endurance, muscle blood flow, and quality of life in older HFpEF patients.

ELIGIBILITY:
Inclusion Criteria for Heart Failure Preserved Ejection Fraction Patients:

* ≥60 years of age, male or female.
* Documented heart failure diagnosis.
* Left ventricular ejection fraction ≥50%.
* Clinically stable (no heart failure hospitalization within prior month).

Inclusion Criteria for Healthy Controls:

* ≥60 years of age, male or female (matched to the age and sex of HFpEF patients).
* No cardiac medications except for statins.
* Sedentary (exercise three days per week or less).

Exclusion Criteria for Heart Failure Preserved Ejection Fraction Patients:

* Greater than moderate valvular disease or congenital heart disease.
* New York Heart Association class IV.
* Any orthopedic or medical condition that would limit exercise testing or training.
* Development of signs and symptoms of myocardial ischemia (1 mm ST segment depression on EKG), or unstable hemodynamics/rhythm, or systolic/diastolic blood pressure >240/110 mmHg during baseline cardiopulmonary (peak VO2) testing.

Exclusion Criteria for Healthy Controls:

* Chronic medical condition (e.g. self reported hypertension, or diabetes, or chronic obstructive pulmonary disease or heart disease)
* Abnormal history or cardiovascular physical exam.
* Segmental wall motion abnormalities or structural valvular abnormalities.
* Left ventricular ejection fraction <50%.
* Any orthopedic or medical condition that would limit exercise testing.
* Development of signs and symptoms of myocardial ischemia (1 mm ST segment depression on EKG), or unstable hemodynamics/rhythm, or systolic/diastolic blood pressure >240/110 mmHg during baseline cardiopulmonary (peak VO2) testing.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-04-17 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Muscle sympathetic nerve activity (MSNA) assessed by direct microneurography | Change from Baseline MSNA at 16 weeks
  Standard microneurographic procedures will be used to directly measure MSNA, at rest and during handgrip exercise and post-exercise cuff occlusion, using the peroneal nerve.

SECONDARY OUTCOMES:
Peak Oxygen Uptake (Peak VO2) assessed by gas exchange indirect calorimetry | Change from Baseline Peak VO2 at 16 weeks.
  Peak VO2 will be measured as the highest oxygen uptake during a peak cycle exercise test on an upright cycle ergometer.
Physical functional performance assessed by Short Physical Performance Battery (SPPB) Test | Change from Baseline physical functional performance at 16 weeks.
  The Short Physical Performance Battery consists of 3 subtasks: standing balance, walking speed, and time to raise from a chair 5 times.
Aerobic endurance assessed by six-minute walk distance | Change from Baseline aerobic endurance at 16 weeks.
  The six-minute walk test is a validated measure of aerobic endurance in patients with heart failure that measures the distance covered in a 6 min period.
Muscle blood flow assessed by brachial artery Doppler Ultrasound | Change from Baseline muscle blood flow at 16 weeks.
  Measurement of brachial artery diameter and blood velocity via Doppler Ultrasound to calculate blood flow.
Quality of life assessed by Kansas City Cardiomyopathy Questionnaire (KCCQ) | Change from Baseline quality of life at 16 weeks.
  The KCCQ is a valid, reliable and responsive health status measure for patients with heart failure.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Haykowsky, PhD, Principal Investigator — University of Texas at Arlington
Locations (1):
- University of Texas at Arlington, Arlington, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abudiab MM, Redfield MM, Melenovsky V, Olson TP, Kass DA, Johnson BD, Borlaug BA. Cardiac output response to exercise in relation to metabolic demand in heart failure with preserved ejection fraction. Eur J Heart Fail. 2013 Jul;15(7):776-85. doi: 10.1093/eurjhf/hft026. Epub 2013 Feb 20. PMID 23426022
- [Background] Bhella PS, Prasad A, Heinicke K, Hastings JL, Arbab-Zadeh A, Adams-Huet B, Pacini EL, Shibata S, Palmer MD, Newcomer BR, Levine BD. Abnormal haemodynamic response to exercise in heart failure with preserved ejection fraction. Eur J Heart Fail. 2011 Dec;13(12):1296-304. doi: 10.1093/eurjhf/hfr133. Epub 2011 Oct 5. PMID 21979991
- [Background] Borlaug BA, Melenovsky V, Russell SD, Kessler K, Pacak K, Becker LC, Kass DA. Impaired chronotropic and vasodilator reserves limit exercise capacity in patients with heart failure and a preserved ejection fraction. Circulation. 2006 Nov 14;114(20):2138-47. doi: 10.1161/CIRCULATIONAHA.106.632745. Epub 2006 Nov 6. PMID 17088459
- [Background] Borlaug BA, Nishimura RA, Sorajja P, Lam CS, Redfield MM. Exercise hemodynamics enhance diagnosis of early heart failure with preserved ejection fraction. Circ Heart Fail. 2010 Sep;3(5):588-95. doi: 10.1161/CIRCHEARTFAILURE.109.930701. Epub 2010 Jun 11. PMID 20543134
- [Background] Borlaug BA, Olson TP, Lam CS, Flood KS, Lerman A, Johnson BD, Redfield MM. Global cardiovascular reserve dysfunction in heart failure with preserved ejection fraction. J Am Coll Cardiol. 2010 Sep 7;56(11):845-54. doi: 10.1016/j.jacc.2010.03.077. PMID 20813282
- [Background] Borlaug BA. The pathophysiology of heart failure with preserved ejection fraction. Nat Rev Cardiol. 2014 Sep;11(9):507-15. doi: 10.1038/nrcardio.2014.83. Epub 2014 Jun 24. PMID 24958077
- [Background] Cleland JG, Tendera M, Adamus J, Freemantle N, Polonski L, Taylor J; PEP-CHF Investigators. The perindopril in elderly people with chronic heart failure (PEP-CHF) study. Eur Heart J. 2006 Oct;27(19):2338-45. doi: 10.1093/eurheartj/ehl250. Epub 2006 Sep 8. PMID 16963472
- [Background] Fisher JP, Young CN, Fadel PJ. Autonomic adjustments to exercise in humans. Compr Physiol. 2015 Apr;5(2):475-512. doi: 10.1002/cphy.c140022. PMID 25880502
- [Background] Gottdiener JS, Arnold AM, Aurigemma GP, Polak JF, Tracy RP, Kitzman DW, Gardin JM, Rutledge JE, Boineau RC. Predictors of congestive heart failure in the elderly: the Cardiovascular Health Study. J Am Coll Cardiol. 2000 May;35(6):1628-37. doi: 10.1016/s0735-1097(00)00582-9. PMID 10807470
- [Background] Granger CB, McMurray JJ, Yusuf S, Held P, Michelson EL, Olofsson B, Ostergren J, Pfeffer MA, Swedberg K; CHARM Investigators and Committees. Effects of candesartan in patients with chronic heart failure and reduced left-ventricular systolic function intolerant to angiotensin-converting-enzyme inhibitors: the CHARM-Alternative trial. Lancet. 2003 Sep 6;362(9386):772-6. doi: 10.1016/S0140-6736(03)14284-5. PMID 13678870
- [Background] Haykowsky MJ, Brubaker PH, John JM, Stewart KP, Morgan TM, Kitzman DW. Determinants of exercise intolerance in elderly heart failure patients with preserved ejection fraction. J Am Coll Cardiol. 2011 Jul 12;58(3):265-74. doi: 10.1016/j.jacc.2011.02.055. PMID 21737017
- [Background] Haykowsky M, Brubaker P, Kitzman D. Role of physical training in heart failure with preserved ejection fraction. Curr Heart Fail Rep. 2012 Jun;9(2):101-6. doi: 10.1007/s11897-012-0087-7. PMID 22430146
- [Background] Haykowsky MJ, Brubaker PH, Morgan TM, Kritchevsky S, Eggebeen J, Kitzman DW. Impaired aerobic capacity and physical functional performance in older heart failure patients with preserved ejection fraction: role of lean body mass. J Gerontol A Biol Sci Med Sci. 2013 Aug;68(8):968-75. doi: 10.1093/gerona/glt011. Epub 2013 Mar 22. PMID 23525477
- [Background] Haykowsky MJ, Kouba EJ, Brubaker PH, Nicklas BJ, Eggebeen J, Kitzman DW. Skeletal muscle composition and its relation to exercise intolerance in older patients with heart failure and preserved ejection fraction. Am J Cardiol. 2014 Apr 1;113(7):1211-6. doi: 10.1016/j.amjcard.2013.12.031. Epub 2014 Jan 15. PMID 24507172
- [Background] Kitzman DW, Little WC, Brubaker PH, Anderson RT, Hundley WG, Marburger CT, Brosnihan B, Morgan TM, Stewart KP. Pathophysiological characterization of isolated diastolic heart failure in comparison to systolic heart failure. JAMA. 2002 Nov 6;288(17):2144-50. doi: 10.1001/jama.288.17.2144. PMID 12413374
- [Background] Kitzman DW, Nicklas B, Kraus WE, Lyles MF, Eggebeen J, Morgan TM, Haykowsky M. Skeletal muscle abnormalities and exercise intolerance in older patients with heart failure and preserved ejection fraction. Am J Physiol Heart Circ Physiol. 2014 May;306(9):H1364-70. doi: 10.1152/ajpheart.00004.2014. Epub 2014 Mar 21. PMID 24658015
- [Background] Liao L, Jollis JG, Anstrom KJ, Whellan DJ, Kitzman DW, Aurigemma GP, Mark DB, Schulman KA, Gottdiener JS. Costs for heart failure with normal vs reduced ejection fraction. Arch Intern Med. 2006 Jan 9;166(1):112-8. doi: 10.1001/archinte.166.1.112. PMID 16401819
- [Background] Massie BM, Carson PE, McMurray JJ, Komajda M, McKelvie R, Zile MR, Anderson S, Donovan M, Iverson E, Staiger C, Ptaszynska A; I-PRESERVE Investigators. Irbesartan in patients with heart failure and preserved ejection fraction. N Engl J Med. 2008 Dec 4;359(23):2456-67. doi: 10.1056/NEJMoa0805450. Epub 2008 Nov 11. PMID 19001508
- [Background] Pitt B, Pfeffer MA, Assmann SF, Boineau R, Anand IS, Claggett B, Clausell N, Desai AS, Diaz R, Fleg JL, Gordeev I, Harty B, Heitner JF, Kenwood CT, Lewis EF, O'Meara E, Probstfield JL, Shaburishvili T, Shah SJ, Solomon SD, Sweitzer NK, Yang S, McKinlay SM; TOPCAT Investigators. Spironolactone for heart failure with preserved ejection fraction. N Engl J Med. 2014 Apr 10;370(15):1383-92. doi: 10.1056/NEJMoa1313731. PMID 24716680
- [Background] Redfield MM. Heart failure--an epidemic of uncertain proportions. N Engl J Med. 2002 Oct 31;347(18):1442-4. doi: 10.1056/NEJMe020115. No abstract available. PMID 12409548
- [Background] Redfield MM. Understanding "diastolic" heart failure. N Engl J Med. 2004 May 6;350(19):1930-1. doi: 10.1056/NEJMp048064. No abstract available. PMID 15128890
- [Background] Shimiaie J, Sherez J, Aviram G, Megidish R, Viskin S, Halkin A, Ingbir M, Nesher N, Biner S, Keren G, Topilsky Y. Determinants of Effort Intolerance in Patients With Heart Failure: Combined Echocardiography and Cardiopulmonary Stress Protocol. JACC Heart Fail. 2015 Oct;3(10):803-14. doi: 10.1016/j.jchf.2015.05.010. PMID 26449998
- [Background] Writing Group Members; Mozaffarian D, Benjamin EJ, Go AS, Arnett DK, Blaha MJ, Cushman M, Das SR, de Ferranti S, Despres JP, Fullerton HJ, Howard VJ, Huffman MD, Isasi CR, Jimenez MC, Judd SE, Kissela BM, Lichtman JH, Lisabeth LD, Liu S, Mackey RH, Magid DJ, McGuire DK, Mohler ER 3rd, Moy CS, Muntner P, Mussolino ME, Nasir K, Neumar RW, Nichol G, Palaniappan L, Pandey DK, Reeves MJ, Rodriguez CJ, Rosamond W, Sorlie PD, Stein J, Towfighi A, Turan TN, Virani SS, Woo D, Yeh RW, Turner MB; American Heart Association Statistics Committee; Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2016 Update: A Report From the American Heart Association. Circulation. 2016 Jan 26;133(4):e38-360. doi: 10.1161/CIR.0000000000000350. Epub 2015 Dec 16. No abstract available. PMID 26673558
- [Background] Yamamoto K, Origasa H, Hori M; J-DHF Investigators. Effects of carvedilol on heart failure with preserved ejection fraction: the Japanese Diastolic Heart Failure Study (J-DHF). Eur J Heart Fail. 2013 Jan;15(1):110-8. doi: 10.1093/eurjhf/hfs141. Epub 2012 Sep 14. PMID 22983988